CLINICAL TRIAL: NCT03653533
Title: Evaluation of the Function "Stop Before Hypoglycemia" on External Insulin Pump Coupled With the Continuous Measurement of Interstitial Glycemia in Type 1 Diabetic Adults
Brief Title: Evaluation of the Function "Stop Before Hypoglycemia" on External Insulin Pump
Acronym: AAHPI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties for recruitment
Sponsor: ARAIR Assistance (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2017-A01988-45
Record Dates: First submitted 2018-06-12; First posted 2018-08-31 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Type I Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MiniMed™ 640G alone (Other): MiniMed™ 640G (insulin pump) is used without Captor CGM Enlite® (captor) at phase 1 and phase 4 of the study. ADDQoL, BIPQ and HADS questionnaire are performed.
  Interventions: Device: MiniMed™ 640G
- MiniMed™ 640G + Captor CGM Enlite® (Other): insulin pump coupled with captor without SmartGuard® function tat phase 2 of the study. ADDQoL, BIPQ and HADS questionnaire are performed.
  Interventions: Device: MiniMed™ 640G; Device: Captor CGM Enlite®
- MiniMed™ 640G + Captor + SmartGuard® (Other): insulin pump + captor + SmartGuard® function are used at phase 3 of the study. ADDQoL, BIPQ and HADS questionnaire are performed.
  Interventions: Device: MiniMed™ 640G; Device: Captor CGM Enlite®; Device: SmartGuard®

INTERVENTIONS:
Device: MiniMed™ 640G — The MiniMed™ 640G corresponds to the medical device = pump using for the delivery of insulin
Device: Captor CGM Enlite® — The Captor CGM Enlite® corresponds to the device added for the measurement of the glycemic level
  Arms: MiniMed™ 640G + Captor + SmartGuard®; MiniMed™ 640G + Captor CGM Enlite®
Device: SmartGuard® — This SmartGuard® function is used to improve the glycemia stability in real condition
  Arms: MiniMed™ 640G + Captor + SmartGuard®

SUMMARY:
This study compares the apparition of hypoglycaemia in type I diabetic patients between 2 phases: the one without the use of SmartGuard® function and the one with the use of SmartGuard® function.

DETAILED DESCRIPTION:
The aim of this study is to compare SmartGuard® function with captor and insulin pump to improve the glycemia stability in real condition.

There are several phases:

* phase 1: insulin pump without captor (12 weeks)
* phase 2: insulin pump with captor and without SmartGuard® function (4X6 days; 4 weeks)
* phase 3: insulin pump with captor and with SmartGuard® function (6X6 days; 6 weeks)
* phase 4: insulin pump without captor (4 weeks)

ELIGIBILITY:
Inclusion Criteria:

* type I diabetic patients undr basal/prandial diet
* treated by insuline
* with no insuline pump during at least 3 months
* with HbA1C dosed during the 3 months before inclusion

Exclusion Criteria:

* minor patients
* pregnant woman
* already participating to another studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2019-10-18 (Actual); Study Completion 2019-10-18 (Actual)

PRIMARY OUTCOMES:
Occurrence of hypoglycemia between a phase with no SmartGuard® function and a phase with SmartGuard® function | 6 days
  The primary outcome is the area between the glycemic curve and the hypoglycemic level (70 mg/dL), measured between the 6 last days of the phase without SmartGuard® function and the 6 last days with the use of SmartGuard® function

CONTACTS AND LOCATIONS:
Locations (1):
- Pole Sante Sud Le Mans, Le Mans, France